CLINICAL TRIAL: NCT06180720
Title: Single-Center, Open, Randomized, Single-Dose, Completely Repeated Crossover Bioequivalence Study to Evaluate the Effects of the Test/Reference Preparation, Entacapone,Levodopa and Carbidopa Tablets (II) in the Postprandial State in Healthy Adult Subjects
Brief Title: Bioequivalence Study of Entacapone,Levodopa and Carbidopa Tablets in the Postprandial State in Healthy Chinese Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Cao Yu, Director of Clinical Trials Center of Affiliated Hospital of Qingdao Universit, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QLG1114-02
Record Dates: First submitted 2023-12-13; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Healthy
MeSH Terms: interventions — entacapone; Levodopa; Carbidopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (T)-Reference (R) (Experimental): In this trial, 36 healthy subjects are planned to be enrolled in fasting. According to the randomization table, subjects will be randomly assigned to the Group A: Test (T)-Reference (R), The washout period (dosing interval) between doses will be at least 2 days. After fasting for at least 10 hours.
  Interventions: Drug: Test (T) Entacapone,Levodopa and Carbidopa Tablets (II); Drug: Reference (R) Entacapone,Levodopa and Carbidopa Tablets (II)
- Reference (R)-Test (T) (Experimental): In this trial, 36 healthy subjects are planned to be enrolled in fasting. According to the randomization table, subjects will be randomly assigned to the Group B: Reference (R)-Test (T), The washout period (dosing interval) between doses will be at least 2 days. After fasting for at least 10 hours.
  Interventions: Drug: Test (T) Entacapone,Levodopa and Carbidopa Tablets (II); Drug: Reference (R) Entacapone,Levodopa and Carbidopa Tablets (II)

INTERVENTIONS:
Drug: Test (T) Entacapone,Levodopa and Carbidopa Tablets (II) — Specification:Levodopa 100mg, Carbidopa 25mg, Entacapone 200mg(Abbreviation: 100mg/25mg/200mg). Produced and supplied by Qilu Pharmaceutical Co.
Drug: Reference (R) Entacapone,Levodopa and Carbidopa Tablets (II) — Specification:Levodopa 100mg, Carbidopa 25mg, Entacapone 200mg(Abbreviation: 100mg/25mg/200mg). Supplied by Qilu Pharmaceutical Co.

SUMMARY:
In this trial, 36 healthy subjects are planned to be enrolled in postprandial, and the postprandial trials will be randomized separately. According to the randomization table, subjects will be randomly assigned to one of the two groups (Group A: TRTR, Group B: RTRT). The washout period (dosing interval) between doses will be at least 2 days. Taking the washout period of 2 days as an example, all subjects will take the corresponding medication according to the randomization table on day 1 of the first cycle trial, day 3 of the second cycle trial, day 5 of the third cycle trial, and day 7 of the fourth cycle trial.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an informed consent form before the trial and fully understand the content, process and possible adverse effects of the trial.
2. Ability to complete research in accordance with the requirements of the pilot program.
3. The subject is willing to be free of pregnancy, sperm or egg donation and to voluntarily use effective contraception from the time of signing (female subject has used effective contraception for 14 days prior to the first dose of the drug) to 6 months after the last dose of the drug.
4. Healthy male and female subjects aged 18 years or older (including 18 years of age).
5. Male subjects weighed no less than 50.0 kg and female subjects weighed no less than 45.0 kg, with a body mass index in the range of 19.0 to 28.0 kg/m2 (including threshold values).

Exclusion Criteria:

1. History of serious medical conditions such as cardiac, hepatic, renal, gastrointestinal, neurological, endocrine, respiratory, and psychiatric abnormalities, which are deemed inappropriate for the participant by the study physician#
2. Abnormalities judged by the clinician to be clinically significant, including physical examination, vital signs examination, electrocardiogram, or clinical laboratory tests#
3. Previous or existing postural hypotension or morning dizziness#
4. Those with bile duct obstruction or a history of bile duct obstruction, or those with narrow-angle glaucoma, chronic open-angle glaucoma, ischemic heart disease, or myocardial infarction disease or history#
5. Previous or existing suspicious and undiagnosed skin lesions or a history of melanoma#
6. Those with a history of malignant nerve blocker syndrome (NMS) and/or non-traumatic rhabdomyolysis#
7. Persons with a history of specific allergies (asthma, etc.) or current allergic diseases (hives, eczema, etc.), or allergies (e.g., persons allergic to two or more medications, foods such as milk, or pollen), or known allergies to carbidopa, levodopa, entacapone, or any of the drug components#
8. Those with dysphagia or any history of gastrointestinal disorders that interfere with drug absorption (e.g., gastric or small bowel resection, atrophic gastritis, peptic ulcer, gastrointestinal bleeding, obstruction, etc.)#
9. Female subjects who are pregnant, breastfeeding, or have a positive pregnancy test result
10. Those who are positive for any one or more of Hepatitis B Surface Antigen, Hepatitis C Antibody, HIV Antibody, or Syphilis Antibody#
11. History of substance abuse within five years, or drug use within three months prior to screening, or positive urine drug screen#
12. Those who consumed an average of more than 14 units of alcohol (1 unit = 360 milliliter of beer or 45 milliliter of spirits with 40% alcohol by volume or 150 milliliter of wine) per week in the 3 months prior to screening, or those who were unable to stop their alcohol intake from 24h prior to dosing until the end of the trial, or those who had a positive breath test for alcohol#
13. Those who smoked an average of more than 5 cigarettes per day in the 3 months prior to screening or those who refused not to use tobacco products during their stay#
14. History of surgical procedure within 3 months prior to screening or planned surgery during the study period#
15. Those who have donated blood or lost a significant amount of blood (>400milliliter, except for physiologic blood loss in females) within 3 months prior to the first dose, or those who have donated ≥2 therapeutic doses of platelets within 1 month#
16. Participation in a clinical trial of any drug and taking the drug within 3 months prior to the first dose#
17. The use of nonselective monoamine oxidase inhibitors (e.g., phenelzine and antiphencyclidine), tricyclic antidepressants, dopamine D2 receptor antagonists (e.g., phenothiazines and risperidone), and isoniazid, phenytoin, and iron salts, metoclopramide, capnography interfering with bile duct excretion, chylomicrons, and small intestinal-glucuronidase (e.g., propoxur and erythromycin), in the 30 days prior to the first dose of the drug, rifampicin and chloramphenicol), pyridoxine, highly protein- bound drugs (e.g., warfarin, salicylic acid, prednisone, and disulfiram), CYP2C9 inhibitors (e.g., amiodarone, cimetidine, isoniazid), and CYP2C9 inducers (e.g., barbiturates, dexamethasone, ritonavir)#
18. Those who received a live attenuated vaccine within 14 days prior to the first dose, or who received a live attenuated vaccine during a planned trial#
19. Those who have taken any prescription medication within 14 days prior to the first dose#
20. Those who have taken any over-the-counter medications, herbs, or supplements within 7 days prior to the first dose#
21. Anyone who has taken a special diet (e.g., grapefruit and products containing grapefruit), or any food or beverage rich in caffeine or xanthines (e.g., coffee, tea, chocolate, cocoa, milk tea, etc.), or who has been subjected to strenuous physical activity, or any other factor that affects the absorption, distribution, metabolism, or excretion of the drug in the 48h prior to the first dose of the drug#
22. Those who have difficulty collecting blood from a vein or have a history of needle and blood sickness#
23. Those who have special dietary requirements or are unable to comply with the uniform rules of the clinical research center#
24. Subjects who are unable to participate in the trial for their own reasons#
25. Subjects judged by other investigators to be unsuitable for participation. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-01-04 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 10hours
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC0-t) | 10hours
  Area under the drug concentration-time curve from time 0 to the last accurately measurable concentration at sample collection time t
Area under the plasma concentration versus time curve (AUC0-∞) | 10hours
  Area Under the Plasma Drug Concentration-Time Curve from Time 0 to Infinite Time

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, Principal Investigator — The Affiliated Hospital of Qingdao University Phase I Clinical Research Center